CLINICAL TRIAL: NCT00878501
Title: A Phase II Randomised, Double-blind, Parallel Group, 4-week Treatment, Adaptive Dose Finding, Multi-centre Study Evaluating the Efficacy, Safety, Tolerability and Pharmacokinetics of up to Three Different Oral Doses of AZD1386 and Placebo in Patients With Osteoarthritis of the Knee
Brief Title: Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of AZD1386 in Patients With Osteoarthritis (OA) of the Knee
Acronym: OA19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after the planned interim analysis.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5090C00019
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: Phase II; Pain
MeSH Terms: conditions — Pain | interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD1386, 90 mg (Experimental)
  Interventions: Drug: AZD1386
- AZD1386, 30 mg (Experimental)
  Interventions: Drug: AZD1386
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — oral, during 4 weeks
  Arms: AZD1386, 90 mg
Drug: AZD1386 — oral, during 4 weeks
  Arms: AZD1386, 30 mg
Drug: Placebo — Oral, during 4 weeks
  Arms: Placebo

SUMMARY:
The primary aim of this study is to investigate if AZD1386 is efficacious as an analgesic in patients with osteoarthritis of the knee and at what dose. This will be done by comparing the effect of AZD1386 to placebo ("inactive substance") on pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OA of the knee
* Male or non pregnant females 40 and 80 years old

Exclusion Criteria:

* A current diagnosis of another form of arthritis, in addition to OA
* History, and/or presence of somatic disease, which may interfere with the objectives

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Leff, MD, Study Director — AZD1386AstraZeneca R&D Wilmington, USA; Ola Svensson, MD, Study Chair — AZD1386AstraZeneca R&D Södertälje, Sweden
Locations (41):
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sofia
- Canada (11):
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Saint Romuald, Quebec
  - Research Site, Sherbrooke, Quebec
- Finland (6):
  - Research Site, Helsinki
  - Research Site, Hyvinkää
  - Research Site, Lahti
  - Research Site, Riihimäki
  - Research Site, Tampere
  - Research Site, Vantaa
- Hungary (6):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Veszprém
- Research Site, Japan, Japan
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Toru
  - Research Site, Warsaw
- Slovakia (8):
  - Research Site, Brastislava
  - Research Site, Komárno
  - Research Site, Liptovský Hrádok
  - Research Site, Poprad
  - Research Site, Považská Bystrica
  - Research Site, Rimavská Sobota
  - Research Site, Žiar nad Hronom
  - Research Site, Žilina

REFERENCES:
- [Derived] Miller F, Bjornsson M, Svensson O, Karlsten R. Experiences with an adaptive design for a dose-finding study in patients with osteoarthritis. Contemp Clin Trials. 2014 Mar;37(2):189-99. doi: 10.1016/j.cct.2013.12.007. Epub 2014 Jan 3. PMID 24394343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International multi-center study, 41sites in North America, Japan and Europe recruited between March and July 2009. 327 participants enrolled into the study
Pre-assignment Details: Patients with past or ongoing intolerability to NSAID´s/COX-2's or paracetamol/acetaminophen or patients with insufficient pain relief from these treatments were included in the study. The WOMAC pain on walking had to be ≥40 mm and ≤90 mm on a Visual Analogue Scale (VAS) at both enrolment and after 1 weeks wash-out of medication (randomisation)
Groups:
- Experimental 90 mg: AZD1386 90 mg twice a day (bid) for 4 weeks
- Experimental 30 mg: AZD1386 30 mg twice a day (bid) for 4 weeks
- Placebo Control: Placebo bid for 4 weeks
Period: Overall Study
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control
Started | 104 (One of these patients did not receive study drug since incorrectly enrolled (mis-randomisation)) | 44 | 93
Interim Analysis | 83 | 37 | 81
Completed | 87 | 37 | 85
Not Completed | 17 | 7 | 8
Not completed — Adverse Event | 11 | 3 | 3
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Incorrect enrolment | 1 | 2 | 0
Not completed — Intake of prohibited concom. medication | 0 | 0 | 1
Not completed — Mis-randomisation of patient | 1 | 0 | 0
Not completed — Administrative | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control | Total
Number analyzed (Participants) | 104 | 44 | 93 | 241
Age Continuous [Median (Full Range); unit: Years]
  median and range | 62 [40 to 79] | 61 [40 to 79] | 61 [40 to 79] | 62 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 32 | 65 | 167
  Male | 34 | 12 | 28 | 74

OUTCOME MEASURES:

1. Primary Outcome: Mean of Week 2 and Week 4 Changes From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain Subscale, 48 Hours Recall.
Description: The WOMAC pain subscale is a self-administered electronic scale with 5 questions (Walking on flat surface, Going up or down stairs, At night while in bed, Sitting or lying, Standing upright). Responses were recorded on a 50-mm line with 100 units. 0 mm indicated no pain and 50 mm indicated extreme pain. The scores were then converted to a 100-mm scale. WOMAC pain was derived by calculating the mean of the VAS scores from the 5 questions with score scale ranging from 0 to 100, 0 being no pain and 100 extreme pain.
Time Frame: Baseline, week 2, week 4.
Population: Number of Participants Analyzed for the stated measure are defined according to the Modified Intention To Treat analysis set whereas numbers provided in the Participant Flow Module correspond to number of participants enrolled.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control
Number analyzed (Participants) | 99 | 42 | 90
mm | -19.05 [-22.89 to -15.21] | -20.05 [-25.75 to -14.34] | -17.54 [-21.55 to -13.52]

2. Secondary Outcome: Mean of Week 2 and Week 4 Changes From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Function Subscale, 48 Hours Recall.
Description: The WOMAC VA 3.1. is a self-administered electronic questionnaire that assesses pain, stiffness and disability related to OA. The Function (daily activities) subscale consists of 17 questions. WOMAC function was derived by calculating the mean of the VAS scores from the 17 questions with scores ranging from 0 to 100, 0 = no difficulty in performing daily activities and 100 = extreme difficulty.
Time Frame: Baseline, Week 2 and Week 4.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control
Number analyzed (Participants) | 99 | 42 | 90
mm | -17.19 [-21.17 to -13.21] | -18.84 [-24.66 to -13.01] | -17.12 [-21.29 to -12.96]

3. Secondary Outcome: Mean of Week 2 and Week 4 Changes From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Stiffness Subscale, 48 Hours Recall.
Description: The WOMAC VA3.1. is a self-administered questionnaire that assesses pain, stiffness and disability related to osteoarthritis. The Stiffness subscale consists of 2 questions (Severity of stiffness after first awakening in the morning and severity of stiffnes after periods of inactivity later in the day). WOMAC stiffness was derived by calculating the mean of the VAS scores from the 2 questions with score scale ranging from 0 to 100, 0 being no stiffness and 100 extreme stiffness.
Time Frame: Baseline, Week 2 and Week 4.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control
Number analyzed (Participants) | 99 | 42 | 90
mm | -16.05 [-20.19 to -11.91] | -17.49 [-23.62 to -11.37] | -17.48 [-21.82 to -13.14]

4. Secondary Outcome: Mean of Week 2 and Week 4 Changes From Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Total Score, 48 Hours Recall
Description: The WOMAC VA3.1. is a self-administered questionnaire that assesses pain, stiffness and disability related to osteoarthritis. It consists of a pain subscale (5 questions), function subscale (17 questions). and a stiffness subscale (2 questions). The total score was derived by calculating the mean of the VAS scores from all 24 questions with score scale ranging from 0 to 100, 0 being no pain, stiffness and difficulty in performing daily activities and 100 being extreme pain, stiffness and difficulty in performing daily activities.
Time Frame: Baseline, Week 2 and Week 4.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control
Number analyzed (Participants) | 99 | 42 | 90
mm | -17.48 [-21.35 to -13.61] | -18.93 [-24.63 to -13.24] | -17.27 [-21.33 to -13.22]

ADVERSE EVENTS:
Description: One participant in the Experimental 90 mg Arm did not receive study drug since incorrectly enrolled and is therefore not included.
Arm/Group | Experimental 90 mg | Experimental 30 mg | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/103 | 1/44 | 1/93
Other Adverse Events (participants affected / at risk) | 61/103 | 15/44 | 14/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental 90 mg (N=103) | Experimental 30 mg (N=44) | Placebo Control (N=93)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental 90 mg (N=103) | Experimental 30 mg (N=44) | Placebo Control (N=93)
Dysgeusia (Nervous system disorders) | 15 | 2 | 1
Hot flush (Vascular disorders) | 8 | 5 | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 10 | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 3 | 0
Feeling cold (General disorders) | 7 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 6 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 4 | 3 | 0
Headache (Nervous system disorders) | 3 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other